CLINICAL TRIAL: NCT04285034
Title: Cardiovascular Function and Ribavirin Pharmacokinetics and Pharmacodynamics in Lassa Fever Patients in Nigeria: a Prospective Observational Cohort Study
Brief Title: Cardiovascular Function and Ribavirin PK/PD in Lassa Fever in Lassa Fever
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: 04-19
Record Dates: First submitted 2020-02-18; First posted 2020-02-26 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: Lassa Fever
MeSH Terms: conditions — Lassa Fever

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — PAXGene (RNA) DBS and FTA cards
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (2):
- Ribavirin only: Patients will receive ribavirin in accordance with Nigerian treatment guidelines. Patients will either receive the McCormick regimen or the Irrua regimen.
  PK blood tests will be done on Day 1,2,5,6,10,11,12,13, discharge; Paxgene RNA blood test on day 1, 3, 5, discharge Haematocrit finger prick test on day 1,2, 5, 6, 10, discharge
- Cardiocascular study only: Cardiac tests (NICAS (daily), ECG (Day 1, 5, 10, discharge), Echocardiogram (Day 1, 5, discharge), Ultrasound (Day 1, 3, 5, 7, 10), Endopat (Day 1 and discharge)) will be done throughout; Haematocrit finger prick test daily PAXgene RNA blood test on day 1, 5, discharge

SUMMARY:
Arenaviruses are included in the World Health Organisation R&D Blueprint list of high priority pathogens, since this virus group includes several epidemic-prone highly pathogenic viruses for which there are inadequate diagnostic, therapeutic, and preventative interventions. Junin, Machupo, Guanarito, Sabia, Lujo, and Lassa virus can all cause a viral haemorrhagic fever with high case fatality in hospitalised cases. Lassa fever is the most common severe arenavirus disease and is endemic across many low and middle income countries in West Africa, with an estimated 37.7 million people in 14 countries living in areas at risk of Lassa virus. Despite the discovery of Lassa virus in 1972 and an estimated 300,000 cases and 5000-10,000 deaths annually, there remain gaps in our understanding of the natural history of disease and in the availability of evidence based interventions.

The protocol has two components. Sites may implement one or both components.

1. Cardiovascular function in Lassa fever: Lassa fever in humans is often described in the literature as being characterized by vascular leak and shock in the terminal phase, this being the main pathway to death. Whilst animal data supports this, there are very limited data in humans. One of the main aims of this study therefore is to characterize cardiovascular function in patients with Lassa fever, with the ultimate goal of informing future trials of supportive or therapeutic strategies to improve vascular leak.
2. Ribavirin pharmacokinetics and pharmacodynamics: The recommended treatment for Lassa is ribavirin, but its efficacy has not been established in randomized controlled trials and its mechanism of action is not fully understood. There are very limited PK data on ribavirin in patients with Lassa fever and the optimal dose of ribavirin for an RCT has not been established. Furthermore, there are various hypothesized mechanisms of action of ribavirin, none of which have been investigated in humans with Lassa fever. Therefore, further aims of this study are to characterize the PK of ribavirin and ribavirin metabolites (RMP, RDP, RTP) in Lassa fever patients and to identify potential mechanisms of action ribavirin in Lassa fever. Understanding Ribavirin's mechanism of action in Lassa fever is important for the optimal design of a future RCT.

DETAILED DESCRIPTION:
Summary of cardiovascular function study Lassa fever carries a treated mortality in hospitalized patients of up to 30%. Lassa fever is often described as being characterized by vascular leak and shock in the terminal phase, but, whilst animal data supports this, there are limited data in humans. A further aim of this study therefore is to characterize cardiovascular function in patients with Lassa fever, with the ultimate goal of informing future trials of supportive or therapeutic strategies.

Summary of ribavirin pharmacokinetics and pharmacodynamics sub-study Lassa fever carries a treated mortality in hospitalized patients of up to 30% in Nigeria. Ribavirin is the current standard of care. However, the efficacy of ribavirin has not been established in RCTs. There is very limited PK data on ribavirin in patients with Lassa fever and the optimal dose of ribavirin for an RCT is unknown. The aim of this study is to characterize the PK of ribavirin in Lassa fever, and identify any associations between ribavirin PK parameters and viral load and markers of inflammatory status.

ELIGIBILITY:
Cardiovascular Study:

Inclusion Criteria:

* Suspected or RT-PCR confirmed Lassa fever diagnosis
* Aged 10 years or above

Exclusion Criteria:

• None

Ribavirin PK/PD study

Inclusion Criteria:

* Suspected or RT-PCR confirmed Lassa fever diagnosis
* Patient will receive ribavirin therapy
* Aged 10 years or above

Exclusion Criteria:

• None

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted to Lassa fever treatment centres with a diagnosis of suspected or RT-PCR confirmed Lassa fever.
Sampling Method: Non-Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2019-11-26 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Cardiovascular | through study completion, an average of 2 weeks
  Mean Arterial Pressure is less than 65mmHg or Systolic Blood Pressure is less than 90mmgHg or pulse pressure < 20mmHg
Ribavirin Pharmacokinetics | through study completion, an average of 2 weeks
  Proportion of patients with ribavirin CMIN above the IC90 at > 80% of measured CMIN during therapy
Ribavirin Pharmacodynamics | 5 days
  Change in Lassa virus Viral Load from baseline to day 5

SECONDARY OUTCOMES:
Cardiovascular | through study completion, an average of 2 weeks
  To identify the frequency of shock
Cardiovascular | through study completion, an average of 2 weeks
  To identify the frequency of persistent shock
Cardiovascular | through study completion, an average of 2 weeks
  To identify the frequency of respiratory distress
Cardiovascular | through study completion, an average of 2 weeks
  To identify the frequency of shock and respiratory distress
Cardiovascular | through study completion, an average of 2 weeks
  To identify the frequency of Death
Ribavirin Pharmacokinetics | through study completion, an average of 2 weeks
  Proportion of patients with ribavirin CMIN above the IC50 at all measured CMIN during therapy
Ribavirin Pharmacokinetics | through study completion, an average of 2 weeks
  Duration of time that ribavirin levels are above the IC90 and IC50
Ribavirin Pharmacokinetics | through study completion, an average of 2 weeks
  Calculation of AUC [AUC∞ and AUCLAST] (ribavirin, ribavirin metabolites)
Ribavirin Pharmacokinetics | through study completion, an average of 2 weeks
  Calculation of CMAX (ribavirin, ribavirin metabolites)
Ribavirin Pharmacokinetics | through study completion, an average of 2 weeks
  Calculation of CMIN (ribavirin, ribavirin metabolites)
Ribavirin Pharmacokinetics | through study completion, an average of 2 weeks
  Calculation of T1/2 (ribavirin, ribavirin metabolites)
Ribavirin Pharmacokinetics | through study completion, an average of 2 weeks
  Volume of distribution (ribavirin, ribavirin metabolites)
Ribavirin Pharmacokinetics | through study completion, an average of 2 weeks
  Calculation of Clearance (ribavirin, ribavirin metabolites)
Ribavirin Pharmacodynamics | 10 days
  Change in Lassa virus Viral Load from baseline to day 3 and day 10
Ribavirin Pharmacodynamics | 10 days
  Change in AST, ALT concentrations from baseline to day 3, 5, 10
Ribavirin Pharmacodynamics | 10 days
  Change in eGFR from baseline to day 3, 5, 10
Ribavirin Pharmacodynamics | 10 days
  Change in Haemoglobin from baseline to day 5, 10
Ribavirin Pharmacodynamics | 5 days
  Change in ISG expression from baseline to day 3, 5
Ribavirin Pharmacodynamics | through study completion, an average of 2 weeks
  Time to negative blood RT-PCR for Lassa virus
Ribavirin Pharmacodynamics | through study completion, an average of 2 weeks
  Requirement for blood transfusion during hospitalisation
Ribavirin Pharmacodynamics | through study completion, an average of 2 weeks
  Reaching KDIGO stage 3 during hospitalisation
Ribavirin Pharmacodynamics | through study completion, an average of 2 weeks
  Requirement for dialysis during hospitalisation
Ribavirin Pharmacodynamics | through study completion, an average of 2 weeks
  Duration of hospitalisation

OTHER OUTCOMES:
Cardiovascular Explanatory | through study completion, an average of 2 weeks
  To identify the frequency of vascular leak
Cardiovascular Explanatory | through study completion, an average of 2 weeks
  To identify the frequency of cardiac function
Cardiovascular Explanatory | through study completion, an average of 2 weeks
  To identify the frequency of total peripheral resistance
Cardiovascular Explanatory | through study completion, an average of 2 weeks
  To identify the frequency of total body water
Cardiovascular Explanatory | through study completion, an average of 2 weeks
  To identify the frequency of Reactive hyperaemic index
Ribavirin Pharmacokinetics Explanatory | through study completion, an average of 2 weeks
  Age
Ribavirin Pharmacokinetics Explanatory | through study completion, an average of 2 weeks
  Gender
Ribavirin Pharmacokinetics Explanatory | through study completion, an average of 2 weeks
  Calculation of eGFR
Ribavirin Pharmacokinetics Explanatory | through study completion, an average of 2 weeks
  Calculation of Total body water
Ribavirin Pharmacokinetics Explanatory | through study completion, an average of 2 weeks
  ITPA, SLC28 gene polymorphisms
Ribavirin Pharmacodynamics Explanatory | through study completion, an average of 2 weeks
  Calculation of AUC [AUC∞ and AUCLAST]
Ribavirin Pharmacodynamics Explanatory | through study completion, an average of 2 weeks
  Calculation of CMAX
Ribavirin Pharmacodynamics Explanatory | through study completion, an average of 2 weeks
  Calculation of CMIN
Ribavirin Pharmacodynamics Explanatory | through study completion, an average of 2 weeks
  ITPA, IL28B and SLC28/29 gene polymorphisms

CONTACTS AND LOCATIONS:
Locations (1):
- Owo Federal Medical Centre, Owo, Ondo State, Nigeria

IPD SHARING:
Plan to Share IPD: No